CLINICAL TRIAL: NCT06365736
Title: The Effect of a Contemplative Nature-based Intervention on Spiritual Well-being: a Randomized Controlled Trial
Brief Title: The Effect of a Contemplative Nature-based Intervention on Spiritual Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Xingjian Ruan, Principal Investigator, University of Twente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240310
Record Dates: First submitted 2024-04-05; First posted 2024-04-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Spiritual Well-being; Healthy
Keywords: nature-based interventions; spiritual well-being; contemplate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contemplative nature intervention (Experimental): Participants will spend 30 minutes in nature per day for 10 times over 14 days. Participants will walk for 10 minutes and then choose a nice spot to sit for 10 minutes. During these minutes they will be asked to be silently present and observe trees, plants, flowers, or other aspects of nature and contemplate their connectedness to nature and their own awareness. Then walk back 10 minutes.
  Interventions: Behavioral: Contemplating in nature

INTERVENTIONS:
Behavioral: Contemplating in nature — Participants will spend 30 minutes in nature per day for 10 times over 14 days.
  Each time, participants will walk for 10 minutes and then choose a nice spot to sit for 10 minutes. During these minutes they will be asked to be silently present and observe trees, plants, flowers or other aspects of nature and contemplate their connectedness to nature and their own awareness. Then walk back 10 minutes.
  Other Names: contemplative nature-based interventions

SUMMARY:
The goal of this randomized control trial is to test if contemplating in nature could benefit spiritual well-being in general adults. The main question it aims to answer is:

Does a 2-week contemplative nature intervention improve spiritual well-being?

Participants in the intervention condition will walk for 10 minutes and then choose a nice spot to sit for 10 minutes. During these minutes they will be asked to be silently present and observe trees, plants, flowers, or other aspects of nature and contemplate their connectedness to nature and their own awareness. Then walk back 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* is 18 years or older;
* has access to a nearby natural environment for walking and sitting activities such as a forest, park, or walking area;
* possesses the physical ability to walk for half an hour;
* has access to a computer or tablet with a stable internet connection and an email address;
* is willing to commit half an hour to engage in nature walks 10 times over 14 days.

Exclusion Criteria:

- NA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Spiritual well-being assessed by Spiritual Attitude and Involvement List Short Form (SAIL-SF) | Change from baseline to post-intervention at 2 weeks.
  On a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), respondents rate in how far they think specific statements about spiritual well-being apply to themselves. Higher scores indicate higher scores of spiritual well-being.
Spiritual well-being assessed by Spiritual Attitude and Involvement List Short Form (SAIL-SF) | Change from Baseline to Short-term follow-up at 1 month.
  On a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), respondents rate in how far they think specific statements about spiritual well-being apply to themselves. Higher scores indicate higher scores of spiritual well-being.
Spiritual well-being assessed by Spiritual Attitude and Involvement List Short Form (SAIL-SF) | Change from baseline to longer-term follow-up at 3 months.
  On a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), respondents rate in how far they think specific statements about spiritual well-being apply to themselves. Higher scores indicate higher scores of spiritual well-being.
Spiritual well-being assessed by Daily Spiritual Experience Scale (DSES) | Change from baseline to post-intervention at 2 weeks.
  The non-theistic items from DSES will be used. Ranging from 1 (multiple times a day) to 6 (never). The item responses were reverse coded prior to analysis so that larger values would reflect a higher level of daily spiritual experiences.
Spiritual well-being assessed by Daily Spiritual Experience Scale (DSES) | Change from baseline to short-term follow-up at 1 month.
  The non-theistic items from DSES will be used. Ranging from 1 (multiple times a day) to 6 (never). The item responses were reverse coded prior to analysis so that larger values would reflect a higher level of daily spiritual experiences.
Spiritual well-being assessed by Daily Spiritual Experience Scale (DSES) | Change from baseline to longer-term follow-up at 3 months.
  The non-theistic items from DSES will be used. Ranging from 1 (multiple times a day) to 6 (never). The item responses were reverse coded prior to analysis so that larger values would reflect a higher level of daily spiritual experiences.

OTHER OUTCOMES:
Client satisfaction of intervention condition assessed by Client Satisfaction Questionnaire (CSQ-8) | From post-intervention to short-term follow-up at 1 month.
  A Likert scale scored from 1 (low satisfaction) to 4 (high satisfaction). Higher score means higher satisfaction with the intervention.
Client satisfaction of active control condition assessed by Client Satisfaction Questionnaire (CSQ-8) | From post-intervention to short-term follow-up at 1 month.
  A Likert scale scored from 1 (low satisfaction) to 4 (high satisfaction). Higher score means higher satisfaction with the intervention.
Client satisfaction of passive control condition assessed by Client Satisfaction Questionnaire (CSQ-8) | From post-intervention to longer term follow-up at 3 months.
  A Likert scale scored from 1 (low satisfaction) to 4 (high satisfaction). Higher score means higher satisfaction with the intervention.
Nature connectedness assessed by Connectedness to Nature Scale (CNS) | Change from baseline to post-intervention at 2 weeks.
  Items are rated on a 5-point scale with endpoints 1 (strongly disagree) and 5 (strongly agree). Higher score means higher sense of oneness with the natural world.
Nature connectedness assessed by Connectedness to Nature Scale (CNS) | Change from baseline to short-term follow-up at 1 month.
  Items are rated on a 5-point scale with endpoints 1 (strongly disagree) and 5 (strongly agree). Higher score means higher sense of oneness with the natural world.
Nature connectedness assessed by Connectedness to Nature Scale (CNS) | Change from baseline to longer-term follow-up at 3 months.
  Items are rated on a 5-point scale with endpoints 1 (strongly disagree) and 5 (strongly agree). Higher score means higher sense of oneness with the natural world.
Nature connectedness assessed by the single item Inclusion of Nature with Self scale (INS) | Change from baseline to post-intervention at 2 weeks.
  Participants were asked to select one of seven different sets of overlapping circles labeled ''self'' and ''nature.'' Scores ranged from 1 (where the circles touched but did not overlap) to 7 (where the two circles entirely overlapped).
Nature connectedness assessed by the single item Inclusion of Nature with Self scale (INS) | Change from baseline to short-term follow-up at 1 month.
  Participants were asked to select one of seven different sets of overlapping circles labeled ''self'' and ''nature.'' Scores ranged from 1 (where the circles touched but did not overlap) to 7 (where the two circles entirely overlapped).
Nature connectedness assessed by the single item Inclusion of Nature with Self scale (INS) | Change from baseline to longer-term follow-up at 3 months.
  Participants were asked to select one of seven different sets of overlapping circles labeled ''self'' and ''nature.'' Scores ranged from 1 (where the circles touched but did not overlap) to 7 (where the two circles entirely overlapped).
Well-being assessed by Mental Health Continuum-Short Form (MHC-SF) | Change from baseline to post-intervention at 2 weeks.
  A 6-point Likert scale scored from "never" to "every day". Higher score means higher level of well-being.
Well-being assessed by Mental Health Continuum-Short Form (MHC-SF) | Change from baseline to short-term follow-up at 1 month.
  A 6-point Likert scale scored from "never" to "every day". Higher score means higher level of well-being.
Well-being assessed by Mental Health Continuum-Short Form (MHC-SF) | Change from baseline to longer-term follow-up at 3 months.
  A 6-point Likert scale scored from "never" to "every day". Higher score means higher level of well-being.
Psychological well-being assessed by Brief INSPIRE-O | Change from baseline to post-intervention at 2 weeks.
  A 5-point Likert scale scored from 0 (not at all) to 4 (a lot). Higher score means higher psychological well-being.
Psychological well-being assessed by Brief INSPIRE-O | Change from baseline to short-term follow-up at 1 month.
  A 5-point Likert scale scored from 0 (not at all) to 4 (a lot). Higher score means higher psychological well-being.
Psychological well-being assessed by Brief INSPIRE-O | Change from baseline to longer-term follow-up at 3 months.
  A 5-point Likert scale scored from 0 (not at all) to 4 (a lot). Higher score means higher psychological well-being.
Stress assessed by Perceived Stress Scale (PSS) | Change from baseline to post-intervention at 2 weeks.
  A 5-point Likert scale scored from 0 (never) to 4 (very often). Higher score means higher level of perceived stress.
Stress assessed by Perceived Stress Scale (PSS) | Change from baseline to short-term follow-up at 1 month.
  A 5-point Likert scale scored from 0 (never) to 4 (very often). Higher score means higher level of perceived stress.
Stress assessed by Perceived Stress Scale (PSS) | Change from baseline to longer-term follow-up at 3 months.
  A 5-point Likert scale scored from 0 (never) to 4 (very often). Higher score means higher level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Bohlmeijer, Prof. Dr., Principal Investigator — University of Twente
Locations (1):
- University of Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No